CLINICAL TRIAL: NCT03856450
Title: Use of Digital Tomosynthesis for Detection and Case Management of Scaphoid and Distal Radius Fractures: A VolumeRAD Data Collection Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 124.02-2018-GES-0001
Record Dates: First submitted 2019-02-01; First posted 2019-02-27 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Distal Radius Fracture; Scaphoid Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Mammography; Diagnostic Imaging; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control-arm group (Active Comparator): The control-arm group will consist of healthy volunteers with no known prior trauma in the wrists. The diagnostic truth for subjects in the control-arm will be no fracture and the treatment truth will be no treatment.
  Interventions: Device: DTS; Device: X-ray
- Test-arm group (Experimental): The test-arm group will consist of subjects who present with a wrist injury and initial SOC X-ray imaging results show a confirmed or suspected distal radius or scaphoid fracture, for which additional diagnostic imaging shall be ordered. Diagnostic truth for subjects in the test-arm will be the per-subject clinical diagnosis and the treatment truth will be the per-subject treatment received.
  Interventions: Device: DTS; Device: X-ray; Device: MRI or CT

INTERVENTIONS:
Device: DTS — Subjects undergo wrist imaging using DTS.
  Other Names: Digital Tomosynthesis (DTS)
Device: X-ray — Subjects undergo wrist imaging using standard X-ray imaging.
  Other Names: X-ray imaging
Device: MRI or CT — Subjects may undergo wrist imaging using MRI or CT.
  Other Names: Magnetic Resonance Imaging (MRI) or Computed Tomography (CT)
  Arms: Test-arm group

SUMMARY:
The study described herein is being conducted to collect clinical data associated with diagnosis and treatment information using the VolumeRAD advanced application.

DETAILED DESCRIPTION:
The study described herein is being conducted to collect clinical data associated with diagnosis and treatment information to support additional, on-label claims for GEHC's VolumeRAD advanced application. The results of this study are intended for use in the submission of FDA 510(k) claims in the United States.

ELIGIBILITY:
Inclusion Criteria for Control-arm Subjects:

Subjects who meet all of the following inclusion criteria may be enrolled in this study:

1. Are adults aged 18 years or older;
2. Are able and willing to comply with study procedures; and
3. Are able and willing to provide written informed consent to participate in this study.

Exclusion Criteria for Control-arm Subjects:

Subjects who meet any of the following exclusion criteria will be excluded from this study:

1. Are documented as pregnant based on PI's medical judgment and in consideration of local clinical practice standards for evidence of pregnancy;
2. Have had known prior trauma in either wrist.

Inclusion Criteria for Test-arm Subjects:

Subjects who meet all of the following inclusion criteria may be enrolled in this study:

1. Are adults aged 18 years or older;
2. Have a confirmed or suspected distal radius or scaphoid wrist fracture;
3. Have completed an X-ray imaging exam per standard of care;
4. Have a standard of care (SOC) CT or MRI exam ordered;
5. Are able and willing to complete DTS imaging exam (if not already completed);
6. Are able and willing to comply with study procedures; and
7. Are able and willing to provide written informed consent to participate in this study.

Exclusion Criteria for Test-arm Subjects:

Subjects who meet any of the following exclusion criteria will be excluded from this study:

1. Are documented as pregnant based on PI's medical judgment and in consideration of local clinical practice standards for evidence of pregnancy;
2. Have additional trauma within the image field of view that either impacts the visualization or changes the treatment of the scaphoid or distal radius fracture;
3. Have had prior reconstructive surgery or fixation in the wrist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of X-ray Images | 1 year
  collection of image sets from X-ray imaging exams for each complete and evaluable subject case
Number of DTS images | 1 year
  Collection of image sets from DTS imaging exams for each complete and evaluable subject case
Number of CT (or MRI) images | 1 year
  collection of image sets from CT (or MRI) imaging exams for each complete and evaluable subject case

SECONDARY OUTCOMES:
Questionnaire about Diagnosis | 1 year
  collection of subject diagnosis (positive, negative, or inconclusive) for each complete and evaluable subject case
Questionnaire about Treatment | 1 year
  collection of treatment information (no treatment necessary, non-operative, operative) for each complete and evaluable subject case

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Hospital - Department of Orthopaedic Surgery, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT03856450/Prot_SAP_000.pdf